CLINICAL TRIAL: NCT01579292
Title: mDPP Pilot RCT of a Motivational Mobile Diabetes Prevention Program (mDPP)
Brief Title: A Mobile Based Diabetes Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1107481
Record Dates: First submitted 2012-04-15; First posted 2012-04-17 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Sedentary Lifestyle; Physical Activity; Pre-Diabetic
MeSH Terms: conditions — Sedentary Behavior; Motor Activity; Glucose Intolerance | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physical Activity and Diet Intervention (Experimental): 5-month physical activity and diet intervention which includes 6 in-person sessions, mobile app, and pedometer
  Interventions: Behavioral: Mobile phone based physical activity with intervention
- Pedometer only (Active Comparator): Pedometer only
  Interventions: Behavioral: Pedometer Only

INTERVENTIONS:
Behavioral: Mobile phone based physical activity with intervention — This group will receive a mobile phone software program and a pedometer. Over a 5-month period, participants in this group will be asked to participate in 6 in-person sessions, wear a pedometer, use a mobile phone physical activity and diet diary, and respond to daily physical activity and diet messages or video clips.
  Arms: Physical Activity and Diet Intervention
Behavioral: Pedometer Only — This group will receive a pedometer. Over a 5-month period, participants in this group will be asked to wear a pedometer.
  Arms: Pedometer only

SUMMARY:
The goals of the study are to:

1. Assess effect sizes of our mDPP intervention on weight loss, physical activity, dietary intake, and fasting plasma glucose (FPG) levels from baseline to 5 months as compared to a control group.
2. To explore the association between low heath-literacy levels at baseline and adherence to mobile phone usage.
3. To conduct process evaluation to gain insights into patient compliance to the mobile intervention, including usage barriers and acceptability of our mDPP, at 1 and 5 months using a semi-structured interview method.

DETAILED DESCRIPTION:
The prevalence of type 2 diabetes (T2DM) continues to rise at an alarming rate in the United States. A greater risk of diabetes is observed for ethnic/racial minority and lower socioeconomic status (SES)groups as compared to Caucasians of similar ages. Several clinical trials have tested intensive lifestyle interventions or pharmacologic agents in preventing or delaying T2DM in adults at risk. These trials (e.g.the Diabetes Prevention Program) consistently show impressive diabetes risk reductions using lifestyle interventions, such as relatively modest amounts of weight loss and exercise. However these programs have been expensive to implement and sustain over time in clinical settings or communities.

Mobile technologies are ideal platforms to deliver and disseminate such lifestyle modification programs to a much broader ethnic/racial minority population, making them more cost effective. Today, 87% of adults in the U.S. own a mobile phone. In particular, usage of non-voice services (such as text messaging or mobile internet) in African-Americans and non-white Hispanics is significantly higher than their Caucasian counterparts. In contrast, ethnic /racial minority populations are much less likely to own a computer at home compared to their Caucasian counterparts. Given the rapid diffusion of mobile technologies in ethnic/racial minority populations, we need to understand how to apply mobile persuasive technologies to such lifestyle modification programs.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary lifestyle at work and/or during leisure time
* Intend to be physically active
* Are over 25 years of age
* Access to a home telephone or a mobile phone
* Speak and read English
* Are not physically active
* Have no disabilities that limit physical activity
* Have high blood sugar (fasting blood sugar 100-125) but do not have diabetes

Exclusion Criteria:

* Known medical conditions or other physical problems that need special attention in an exercise program
* Plan a trip abroad during the first 5 months of the study period.
* Pregnant/Delivered a baby during the last 6 months
* Known severe hearing or speech problem
* Currently participate in lifestyle modification programs or research studies that may potentially confound the results of the study
* History of gastric bypass surgery or future plans for gastric bypass surgery in the next 5 months
* Already taking medication for diabetes
* Recovery from addiction
* Known eating disorders
* Bmi over 25 if non-Asian or over 23 if Asian

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2012-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Body weight (kg) | 5 months
Body mass index | 5 months

SECONDARY OUTCOMES:
Physical activity measured by Omron Active Style Pro HJA-350IT pedometer | 5 months
Total daily calories (kcal) | 5 months
Daily calories from fat (kcal) | 5 months
Fasting plasma glucose | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Yoshimi Fukuoka, Ph.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States